CLINICAL TRIAL: NCT03408782
Title: The Association of Surgical Drains With the Risk of Surgical Site Infection - a Prospective Observational Study
Brief Title: Drains and Surgical Site Infections
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Edin Mujagic, Edin Mujagic, MD, University Hospital, Basel, Switzerland
Other Study IDs: ch10Weber
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Surgical Site Infection
Keywords: Surgical Site Infection; Surgical drains
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No drainage: Those patients that underwent surgery and no drain was inserted at the end of the procedure
- Drainage: Those patients that underwent surgery and one or several drains were inserted at the end of the procedure.
  Interventions: Procedure: Insertion of drainage

INTERVENTIONS:
Procedure: Insertion of drainage
  Groups: Drainage

SUMMARY:
This prospective observational study examines the associations of presence, duration, type, number and location of surgical drains with the risk of surgical site infections in a contemporary and multicentric cohort of general, orthopedic trauma and vascular surgery procedures.

DETAILED DESCRIPTION:
Surgical site infections (SSI) represent the most common type of nosocomial infection amongst surgical patients. They cause morbidity and mortality.

Surgical Drains are commonly inserted at the end of many surgical procedures. In contrast to potential benefits, drains are also thought to potentially serve as a conduit of bacteria into the wound and hence may increase the risk of SSI. Patterns of use of drains vary widely across surgical disciplines and individual practices. There are no uniform guidelines and standards are often rather based on tradition than on evidence. The aim of this large prospective study was to examine the association of presence, duration, type, number and location of drains with the risk of SSI in a contemporary and multicentric cohort of general, orthopedic trauma and vascular surgery procedures.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients
* Age 18 years or older
* General, orthopedic trauma and vascular procedures
* Surgical antimicrobial prophylaxis

Exclusion Criteria:

* outpatient surgery
* Presence of a contraindication for cefuroxime and/or metronidazole
* preexisting antibiotic therapy within 14 days prior to surgery
* cognitive impairment
* combined operations including other than the above specified surgical divisions
* Emergency procedures with planned incision within 2 hours after indicating the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study is nested in a multicenter randomized controlled trial that was designed to evaluate the optimal timing of surgical antimicrobial prophylaxis in a general, orthopedic trauma and vascular surgery population. The term "general surgery" refers to gastrointestinal, oncologic breast, endocrine and hernia surgery. The study centers are two tertiarry referral hospitals in Switzerland. All patients included in the randomized controlled trial are included in this observational study as well.
Sampling Method: Probability Sample
Enrollment: 4584 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days
  The occurrence of surgical site infection according to CDC criteria

CONTACTS AND LOCATIONS:
Overall Officials: Edin Mujagic, MD, Principal Investigator — University Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weber WP, Mujagic E, Zwahlen M, Bundi M, Hoffmann H, Soysal SD, Kraljevic M, Delko T, von Strauss M, Iselin L, Da Silva RXS, Zeindler J, Rosenthal R, Misteli H, Kindler C, Muller P, Saccilotto R, Lugli AK, Kaufmann M, Gurke L, von Holzen U, Oertli D, Bucheli-Laffer E, Landin J, Widmer AF, Fux CA, Marti WR. Timing of surgical antimicrobial prophylaxis: a phase 3 randomised controlled trial. Lancet Infect Dis. 2017 Jun;17(6):605-614. doi: 10.1016/S1473-3099(17)30176-7. Epub 2017 Apr 3. PMID 28385346
- [Background] Mujagic E, Zwimpfer T, Marti WR, Zwahlen M, Hoffmann H, Kindler C, Fux C, Misteli H, Iselin L, Lugli AK, Nebiker CA, von Holzen U, Vinzens F, von Strauss M, Reck S, Kraljevic M, Widmer AF, Oertli D, Rosenthal R, Weber WP. Evaluating the optimal timing of surgical antimicrobial prophylaxis: study protocol for a randomized controlled trial. Trials. 2014 May 24;15:188. doi: 10.1186/1745-6215-15-188. PMID 24885132